CLINICAL TRIAL: NCT06694324
Title: Liposomal Doxorubicin Hydrochloride and Apatinib in Combination with Camrelizumab for the First-line Treatment of Advanced/unresectable Dedifferentiated Liposarcoma
Brief Title: First-line Treatment of Advanced/unresectable DDLPS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhiguo Luo, MD, PhD, Chief Clinical Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fudan-CMS-001
Record Dates: First submitted 2024-11-12; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-09

CONDITIONS: Dedifferentiated Liposarcoma; Soft Tissue Sarcoma (STS)
Keywords: liposomal doxorubicin; apatinib; Camrelizumab; first line treatment
MeSH Terms: conditions — Liposarcoma; Sarcoma | interventions — liposomal doxorubicin; apatinib; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Liposomal Doxorubicin+Apatinib+Camrelizumab (Experimental): The patients with advanced or unresectable de-differentiated liposarcoma will be enrolled and given Liposomal doxorubicin hydrochloride: 30 mg/m2, d1, IV over 30 min; apatinib: 250 mg, qd; and karelizumab: 200 mg, d1, IV; Q3W, continued treatment for 6 cycles followed by apatinib and camrelizumab until disease progression, development of unacceptable toxicity, or death of the patient or 2 years of treatment.
  Interventions: Drug: Liposomal Doxorubicin (Doxil); Drug: Apatinib; Drug: Camrelizumab

INTERVENTIONS:
Drug: Liposomal Doxorubicin (Doxil) — 30 mg/m2, d1, IV
Drug: Apatinib — 250 mg, qd
Drug: Camrelizumab — 200 mg, d1, IV

SUMMARY:
Evaluating the efficacy and safety of liposomal doxorubicin hydrochloride and apatinib in combination with camrelizumab for the first-line treatment of advanced/unresectable dedifferentiated liposarcoma

DETAILED DESCRIPTION:
Based on the clinical benefits provided by doxorubicin liposome, apatinib and camrelizumab treatment in STS, this study intends to explore the efficacy and safety of doxorubicin liposome hydrochloride and apatinib combined with camrelizumab in the first-line treatment of advanced/unresectable dedifferentiated liposarcoma with the aim of providing a better therapeutic option for the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years, male or female;
2. Histologically confirmed dedifferentiated liposarcoma;
3. metastatic stage not having received systemic therapy;
4. no brain metastases;
5. ECOG PS: 0~1 points;
6. normal function of major organs, meeting the following requirements (within 7 days prior to initiation of study treatment): 1)Left ventricular ejection fraction (LVEF) ≥50%; 2)Normal electrocardiogram; 3)Hemoglobin [HB] ≥ 90 g/L; 4)Absolute neutrophil count [ANC] ≥1.5×109/L; 5) Platelet [PLT] ≥100×109/L; 6)Serum total bilirubin [TBIL] ≤1.5 times the upper limit of normal (ULN); 7) alanine aminotransferase [ALT], aspartate aminotransferase [AST] <2.5 × ULN; if there are liver metastases, ALT and AST ≤5 × ULN; 8) Serum creatinine [Cr] ≤ 1 × ULN or endogenous creatinine clearance > 50 ml/min (Cockcroft-Gault formula);
7. women of childbearing potential must have a negative pregnancy test (serum or urine) within 7 days prior to enrollment and voluntarily use an appropriate method of contraception for the duration of the observation period and for 8 weeks after the final administration of study drug; in the case of males, they should be surgically sterilized or agree to use an appropriate method of contraception for the duration of the observation period and for 8 weeks after the final administration of study drug;
8. expected to have good compliance and be able to follow up on efficacy and adverse effects as required by the protocol;
9. sign an informed consent form.

Exclusion Criteria:

1. patients with recurrence within six months of postoperative adjuvant therapy;
2. previous adjuvant or neoadjuvant phase with cumulative dose of doxorubicin, liposomal doxorubicin, or other anthracyclines ≥ 240 mg/m2;
3. Use of PD-1 or PD-L1 inhibitors in prior adjuvant or neoadjuvant phase;
4. patients with prior adjuvant or neoadjuvant phase use of apatinib mesylate and patients with prior treatment with vascular endothelial growth inhibitor-targeted agents such as sunitinib, sorafenib, bevacizumab, imatinib, famitinib, pazopanib, regorafenib, and erlotinib.
5. Other active malignancies within 5 years or concurrently;
6. central nervous system involvement;
7. clinical symptoms or diseases of the heart that are not well controlled, such as (1) cardiac insufficiency of grade II or higher according to the New York Heart Association (NYHA) criteria or cardiac ultrasound: LVEF (Left Ventricular Ejection Fraction) < 50%; (2) unstable angina pectoris; (3) myocardial infarction within 1 year prior to the start of study treatment; (4) clinically significant supraventricular or ventricular arrhythmia Need for treatment or intervention: (5) QTc >450 ms (men); QTc >470 ms (women) (QTc intervals are calculated using the Fridericia formula; if the QTc is abnormal, three consecutive measurements may be taken at approximately 2-minute intervals and averaged);
8. patients with signs or history of bleeding, regardless of severity; any bleeding or bleeding event CTCAE grade 3 within 4 weeks prior to enrollment, unhealed wounds, ulcers, or fractures
9. those with hypertension that cannot be reduced to the normal range (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg) with antihypertensive medication (based on the average of BP readings obtained from ≥2 measurements) are permitted to achieve the above parameters with the use of antihypertensive therapy;
10. patients with severe hepatic or renal insufficiency (grade 4);
11. poorly controlled diabetes mellitus (FBG) > 10 mmol/L);
12. Patients with active ulcers, intestinal perforation, intestinal obstruction;
13. Routine urinalysis showing urinary protein++, confirming 24-hour urine protein quantification >1.0g;
14. Presence of active autoimmune disease or history of autoimmune disease with possible relapse;
15. Uncontrolled infection or unexplained fever >38.5°C at screening;
16. a known history of severe allergy to the study drug;
17. other patients deemed unsuitable for inclusion by the treating physician.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
overall response rate, ORR | up to two years
  the best response rate

SECONDARY OUTCOMES:
progression free survival, PFS | up to three years
  from first dose treatment to disease progression
overall survival, OS | up to three years
  overall survival
adverse events, AE | up to three years
  treatment related adverse events, TRAEs

CONTACTS AND LOCATIONS:
Overall Officials: Zhiguo Luo, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University, Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
The researchers decided not to share